CLINICAL TRIAL: NCT00487656
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase-2B Study to Assess the Safety and Efficacy Effects of ART-123 on Subjects With Sepsis and Disseminated Intravascular Coagulation
Brief Title: Safety and Efficacy of ART-123 in Subjects With Sepsis and Disseminated Intravascular Coagulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Artisan Pharma, Inc. (Industry)
Responsible Party: Inder Kaul, Chief Medical Officer, Artisan Pharma, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-001; NCT01090115 (obsolete NCT alias)
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Sepsis; Disseminated Intravascular Coagulation
MeSH Terms: conditions — Sepsis; Disseminated Intravascular Coagulation | interventions — ART123

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ART-123 (Experimental): 6 mg/ml ampule solution for injection
  Interventions: Drug: ART-123
- Placebo (Placebo Comparator): 6 mg/mlampule of solution for injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ART-123 — 6mg/ml ampule solution for injection @ .01mg/kg
  Arms: ART-123
Drug: placebo — 6 mg/ml ampule solution for injection at .01mg/kg
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if ART-123 (recombinant human soluble thrombomodulin) decreases the number of people who die as a result of Disseminated Intravascular Coagulation (DIC) complication of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Infection or suspected infection resulting in sepsis and DIC

Exclusion Criteria:

* Unable to provide informed consent, or lack of consent from an acceptable surrogate
* Subjects < 18 years of age
* Known conditions that could confound the diagnosis of DIC due to sepsis
* Known conditions that increase the risk of bleeding
* Known medical condition associated with a hypercoagulable state
* Known or suspected severe liver disease
* History of solid organ (excluding uncomplicated kidney), bone marrow or stem cell transplantation
* Renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2007-07; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
28-Day All-cause mortality | 28 day

CONTACTS AND LOCATIONS:
Locations (62):
- United States (49):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tuscon, Arizona
  - Bakersfield, California
  - Colton, California
  - Loma Linda, California
  - Long Beach, California
  - Los Angeles, California
  - Rancho Mirage, California
  - San Diego, California
  - San Francisco, California
  - Stanford, California
  - Hartford, Connecticut
  - Bay Pines, Florida
  - Celebration, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Springfield, Illinois
  - Kansas City, Kansas
  - Topeka, Kansas
  - Hazard, Kentucky
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Springfield, Massachusetts
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Pontiac, Michigan
  - Camden, New Jersey
  - Englewood, New Jersey
  - Newark, New Jersey
  - Flushing, New York
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Toledo, Ohio
  - Danville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Knoxville, Tennessee
  - Houston, Texas
  - Lackland Air Force Base, Texas
- Canada (8):
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Kingston, Ontario
  - London, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Windsor, Ontario
  - Greenfield Park, Quebec
- Malaysia (3):
  - Kuala Pahang
  - Lumpur
  - Sarawak
- Thailand (2):
  - Chiang Mai
  - Nakhonratchasima